CLINICAL TRIAL: NCT00465036
Title: Effect of Whole Flaxseeds and Flaxseed Mucilage on Lipid Absorption, Glucose and Insulin Metabolism and Appetite Regulation
Brief Title: Effect of Flaxseed on Lipid Uptake and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: KF 01 309595; B226
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Obesity
Keywords: fat absorption; fibres
MeSH Terms: conditions — Obesity | interventions — (1-6)-alpha-glucomannan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Whole flaxseeds, flaxseed mucilage, glucomannan

SUMMARY:
Randomized trial to test the effect of flaxseed fractions on appetite regulation and intestinal lipid absorption.

DETAILED DESCRIPTION:
Randomized multiple crossover trial in 18 healthy males aged 18 to 40 years each are required to complete a total of five iso-caloric meal tests lasting approximately 8½ hours. Test meals will be given as breakfast meals, in which different fractions of flaxseeds are incorporated into baked products. Appetite will be registered using visual analogue scales during 7 hours after the test meal and a total of 10 blood samples will be drawn to evaluate TAG in chylomicrons, plasma LDL, HDL and total cholesterol, plasma TAG, insulin, glucose and appetite hormone levels. At the end of the test day an ad libitum meal will be served and food intake registered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18-40 years
* Normal weight or moderately overweigh (BMI 25-30 kg/m2)

Exclusion Criteria:

* Blood drawing/donation less than six months prior to start of the study
* Hemoglobin concentration <8mmol/L
* Chronic diseases (i.e. diabetes, CVD), hypertension, hyperlipidemia
* Consumption of dietary supplements including vitamin tablets
* Smoking
* Excess physical activity (>10h of intense physical activity per week)
* Medicine use (not including occasional consumption of pain killers)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2006-10; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
TAG in chylomicrons
serum TAG
HDL, LDL and total cholesterol
appetite scores
ad libium food intake
appetite hormone levels

SECONDARY OUTCOMES:
free fatty acid profile
plasma glucose
plasma insulin
meal macronutrient composition
meal energy content
meal pleasantness

CONTACTS AND LOCATIONS:
Overall Officials: Søren Toubro, MD, Principal Investigator — Institute of Human Nutrition
Locations (1):
- Institute of Human Nutrition, Frederiksberg C, Denmark